CLINICAL TRIAL: NCT00345098
Title: A Double-Blind, Multi-Center, Multinational, Randomized Withdrawal Study Evaluating the Efficacy and Safety of SR58611A (350mg q12) Versus Placebo in the Prevention of Depression Relapse up to 1 Year in Patients With Major Depressive Disorder Improved After 12 Weeks of Open Treatment With SR58611A (350mg q12)
Brief Title: A Study of SR58611A in the Prevention of Depression Relapse in Patients With Major Depressive Disorder
Acronym: CALYPSO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LTE5376; EudraCT 2005-004006-81
Record Dates: First submitted 2006-06-26; First posted 2006-06-27 (Estimated); Last update posted 2009-03-12 (Estimated); Status verified 2009-03

CONDITIONS: Depressive Disorder; Major Depression
Keywords: Depression, Antidepressive agents; Clinical Trial; Phase III; Multicenter study
MeSH Terms: conditions — Depressive Disorder; Depressive Disorder, Major; Depression | interventions — Amibegron hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: SR58611A

SUMMARY:
The purpose of the study is to assess whether treatment with SR58611A can prevent relapse of depressive symptoms in patients with major depressive disorder. Relapse will be assessed using the MADRS scale.Patients who demonstrate improvement in depressive symptoms at the end of the initial 12-week open-label treatment period with SR58611A are randomized to continue SR58611A or switch to placebo under double blind conditions for up to 52 weeks of additional treatment. The secondary objective is to evaluate the safety of SR58611A in patients with MDD.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Major Depressive Disorder, Recurrent according to DSM-IV-TR criteria Diagnostic and Statistical Manual of Mental Disorders (Fourth Edition) and assessed with the Mini International Neuropsychiatric Interview (MINI)
* Total score on the Montgomery and Asberg Depression Rating Scale (MADRS) > 28
* At W12 (V7), patients will be randomized into the double-blind treatment phase if they have MADRS total score < 12

Exclusion Criteria:

* Patients with a significant risk of suicide.
* Patients whose current depressive episode is diagnosed with psychotic features, catatonic features, seasonal pattern or post-partum onset.
* Patients with a current depressive episode secondary to a general medical disorder.
* Patients with a lifetime history or presence of bipolar disorder, psychotic disorder, panic disorder and antisocial personality disorder.
* Patients with severe or unstable concomitant medical conditions
* Patients with clinically significant abnormal laboratory value at screening
* The investigator will evaluate whether there are other reasons why a patient may not participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 704 (Actual)
Dates: Start 2006-05; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is the time to relapse of depressive symptoms (in days) during the double-blind study phase.

SECONDARY OUTCOMES:
Change in Clinical Global Impression Severity score. Change in MADRS total score. Change in HAM-A total score

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (13):
- Sanofi-Aventis Administrative Office, Buenos Aires, Argentina
- Sanofi-Aventis Administrative Office, Sofia, Bulgaria
- Sanofi-Aventis Administrative Office, Zagreb, Croatia
- Sanofi-Aventis Administrative Office, Prague, Czechia
- Sanofi-Aventis Administrative Office, Helsinki, Finland
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, México, Mexico
- Sanofi-Aventis Administrative Office, Warsaw, Poland
- Sanofi-Aventis Administrative Office, Bucharest, Romania
- Sanofi-Aventis Administrative Office, Moscow, Russia
- Sanofi-Aventis Administrative Office, Belgrade, Serbia
- Sanofi-Aventis Administrative Office, Bratislava, Slovakia
- Sanofi-Aventis Administrative Office, Midrand, South Africa

REFERENCES:
- See also: Related Info — http://www.sanofi-aventis.com